CLINICAL TRIAL: NCT04182243
Title: Job Satisfaction of Emergency Ambulance Personnel in Northern Cyprus
Brief Title: Job Satisfaction of Emergency Ambulance Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Semra Aslay, Ass. Prof. (M.D.), European University of Lefke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Job Satisfaction
Record Dates: First submitted 2019-11-21; First posted 2019-12-02 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Job Stress
Keywords: Job Satisfaction; Emergency Health Care; Paramedic; Emergency Medical Technician; Nurse
MeSH Terms: conditions — Occupational Stress | interventions — Association

STUDY DESIGN:
Intervention Model Description: The research is a descriptive study to evaluate the working conditions and job satisfaction of nurses, paramedics, and EMTs working in Northern Cyprus. There are 138 nurses, paramedics, and EMTs working in 112 ambulance services. In the research, a complete census conducted without any sampling, and 132 staff interviewed. Four of the six nurses who were not interviewed were on long-term leave and were not on duty at the time of the study. Two nurses who were not included in the survey stated that they did not agree to participate in the study. The researcher conducted the study by appointment in the work environment between October 20 - November 10, 2016, to the health personnel participants working in 112 Emergency Departments of the Ministry of Health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency Health Care Provider (Other): Working in emergency health services in Northern Cyprus
  Interventions: Other: Evaluation of job satisfaction in emergency health care providers by questionnaire

INTERVENTIONS:
Other: Evaluation of job satisfaction in emergency health care providers by questionnaire
  Other Names: Nature of work; Relations with co-workers; Vocational training; Relationship with supervisors; Economic aspect; Cultural aspect; Social aspect; Capacity of consumables

SUMMARY:
The emergency department crowding is a worldwide health problem. Overcapacity admissions result in a decrease in health care quality. High job satisfaction, proper working environment, appropriate institutional structuring in government, and sufficient resources of the staff mean the quality of health care. To evaluate the job satisfaction of the personnel works in emergency health care in North Cyprus and contribute to raising the quality of health services to world standards. In this study, job satisfaction of the personnel working in emergency health services in North Cyprus evaluated through a questionnaire made between October 20; November 10, 2016. It consisted of two parts in which sociodemographic characteristics and job satisfaction scale. The job satisfaction scale developed by Güneri (2011) was a 5-point Likert type. It consisted of 7 sub-dimensions: the nature of work, relations with co-workers, vocational training, relationships with supervisors, economic, cultural, social aspect, and capacity of consumables. The scale can have the lowest score of 47 and the highest score of 235. Participants' high scores on the scale indicated high job satisfaction. The participants', 31.82% were in the 36-49 age, 81.06% were women, 75% were married, 82.5% had children, and 42.42% was an undergraduate degree. The majority of the participants were nurses who had been working for more than ten years and 40-50 hours per week. No significant difference found between job satisfaction and sociodemographic characteristics (p>0.05). High school graduates, head nurses, emergency call center staff, working 1-4 years, 40-50 hours per week, and those who received updating training have significantly higher job-satisfaction scores than the other groups (p<0.05). The high job satisfaction of the personnel working in emergency health services is the meaning of high-quality health care. We recommend the inclusion of emergency health services in the existing structure of the Ministry of Health in Northern Cyprus. Also, emergency health care should be provided by paramedics and EMTs (Emergency Medical Technician), decreasing weekly working hours and increasing updating training.

DETAILED DESCRIPTION:
Perception and evaluation of the environment, communication, comfort, and adaptation to conditions affect individual success in the workplace. Wages and working hours, type of contract (shift work, overtime), security, administration, and relations with co-workers are examples of these conditions. For having high job satisfaction, it is also essential that the staff has sufficient knowledge about the job and their expectations. Job satisfaction can be positively affected by determining job, working time, and eliminating differences of work conditions to emergency health care personnel, especially paramedics.

Emergency health services are not a separate unit in the ministry of health in Northern Cyprus. Since the emergency health services are not directly different from the existing system, and therefore, the staff directly connect to their units, some of the participants work in health centers. The first recruitment as a paramedic in Northern Cyprus in the Ministry of Health took place in 2005. However, Paramedics and EMTs who participated in our study declared that they work under the name of nurse staff. Paramedics, who previously worked under the name of another status, first started to work in the public sector in their occupation group as of 2018. Therefore, the current statistical information of both the ministry of health and the most crowded public hospital in Northern Cyprus does not provide sufficient up-to-date information on the number of paramedics and EMTs.

This descriptive study was conducted to evaluate job satisfaction of nurses, paramedics, and EMTs working in Northern Cyprus emergency health care. A total of 17 healthcare facilities providing emergency care services were in the study. Of these facilities, 2 are emergency call centers, 4 are hospital emergency services, and the rest of connected to health centers. A total of one head nurse, 123 nurses, 12 paramedics, and 3 EMTs provide emergency health care to all of Northern Cyprus.

The data of the study collected between October 20; November 10, 2016, after obtaining permission from the related institutions. The questionnaire consisted of two parts with sociodemographic characteristics and job satisfaction scale. The job satisfaction scale developed by Güneri, İlhan& Avcı was a 5-point Likert type. It consisted of 7 sub-dimensions: the nature of work, relations with co-workers, vocational training, relationships with supervisors, economic, cultural, social aspect, and capacity of consumables.

The answers to suggestions in the scale were scored as "very satisfied = 5 points", "satisfied = 4 points", "okay= 3 points", "dissatisfied = 2 points", and "very dissatisfied = 1 point". The scale lowest score was 47, and the highest was 235. Participants' high scores on the scale indicated high job satisfaction. In this study, the Cronbach alpha coefficient was found to be 0.94 in the scale and 0.79-0.95 in the sub-dimensions.

For statistical analysis, we used to statistical program SPSS 21.0. (SPSS Inc, Chicago, IL, USA). Before the data analysis, the data set checked to eliminate the errors that may arise from data entry. Frequency analysis was used to determine the sociodemographic characteristics of the participants. Scores obtained from job satisfaction scale and sub-dimensions gave as descriptive statistics for central tendency measures such as mean, standard deviation, minimum, and maximum value. The scores of the participants obtained from the job satisfaction scale according to their independent variables were analyzed. For the data analyzing, the Kolmogorov-Smirnov test and the QQ plot graph used. It concluded that the data set conforms to normal distribution. After that, we compared the scale scores according to independent variables.

In the comparison of job satisfaction scores according to the characteristics of the participants such as gender and marital status, a t-test was used since the independent variable consists of two categories. ANOVA test was used to compare the scores obtained by the participants if the independent variable such as age group and professional seniority consisted of more than two categories. If there was a difference between the types of the independent variable as a result of ANOVA, Tukey test was used to determine which groups the dispute originated. In this study, 132 of 138 personnel working in emergency health services reached in Northern Cyprus. Of the remaining, four were on long-term leave, and two did not accept.

ELIGIBILITY:
Inclusion Criteria:A total of 17 healthcare facilities providing emergency care services were in the study.

Exclusion Criteria:

Doctors, did not accept to join to study, long term leaving from job

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Job Satisfaction of Emergency Health Care Providers in Northern Cyprus | Through study completion, an average of 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Semra Aslay, MD, Study Director — European University of Lefke

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participating data
Supporting Information: SAP
Time Frame: After published there is no ending time frame
Access Criteria: Paramedic, EMT, and nurses in emergency health care in Northern Cyprus included in the study. In the research, a complete census conducted without any sampling, and 132 staff interviewed.

REFERENCES:
- [Result] Coomber B, Barriball KL. Impact of job satisfaction components on intent to leave and turnover for hospital-based nurses: a review of the research literature. Int J Nurs Stud. 2007 Feb;44(2):297-314. doi: 10.1016/j.ijnurstu.2006.02.004. Epub 2006 Apr 24. PMID 16631760
- [Result] Gedif G, Sisay Y, Alebel A, Belay YA. Level of job satisfaction and associated factors among health care professionals working at University of Gondar Referral Hospital, Northwest Ethiopia: a cross-sectional study. BMC Res Notes. 2018 Nov 20;11(1):824. doi: 10.1186/s13104-018-3918-0. PMID 30458846
- [Result] Golbasi Z, Kelleci M, Dogan S. Relationships between coping strategies, individual characteristics and job satisfaction in a sample of hospital nurses: cross-sectional questionnaire survey. Int J Nurs Stud. 2008 Dec;45(12):1800-6. doi: 10.1016/j.ijnurstu.2008.06.009. Epub 2008 Aug 13. PMID 18703192
- [Result] Lu H, Barriball KL, Zhang X, While AE. Job satisfaction among hospital nurses revisited: a systematic review. Int J Nurs Stud. 2012 Aug;49(8):1017-38. doi: 10.1016/j.ijnurstu.2011.11.009. Epub 2011 Dec 19. PMID 22189097
- [Result] Ozturk H, Babacan E. The occupational safety of health professionals working at community and family health centers. Iran Red Crescent Med J. 2014 Oct 5;16(10):e16319. doi: 10.5812/ircmj.16319. eCollection 2014 Oct. PMID 25558383
- [Result] Reichard AA, Marsh SM, Tonozzi TR, Konda S, Gormley MA. Occupational Injuries and Exposures among Emergency Medical Services Workers. Prehosp Emerg Care. 2017 Jul-Aug;21(4):420-431. doi: 10.1080/10903127.2016.1274350. Epub 2017 Jan 25. PMID 28121261
- [Result] Maguire BJ. Violence against ambulance personnel: a retrospective cohort study of national data from Safe Work Australia. Public Health Res Pract. 2018 Mar 15;28(1):28011805. doi: 10.17061/phrp28011805. PMID 29582039
- [Result] Sveinsdottir H, Biering P, Ramel A. Occupational stress, job satisfaction, and working environment among Icelandic nurses: a cross-sectional questionnaire survey. Int J Nurs Stud. 2006 Sep;43(7):875-89. doi: 10.1016/j.ijnurstu.2005.11.002. Epub 2005 Dec 19. PMID 16360157
- [Result] Tarcan M, Hikmet N, Schooley B, Top M, Tarcan GY. An analysis of the relationship between burnout, socio-demographic and workplace factors and job satisfaction among emergency department health professionals. Appl Nurs Res. 2017 Apr;34:40-47. doi: 10.1016/j.apnr.2017.02.011. Epub 2017 Feb 3. PMID 28342622
- [Result] Tavakoli N, Shaker SH, Soltani S, Abbasi M, Amini M, Tahmasebi A, Hosseini Kasnavieh SM. Job Burnout, Stress, and Satisfaction among Emergency Nursing Staff after Health System Transformation Plan in Iran. Emerg (Tehran). 2018;6(1):e41. Epub 2018 Jul 13. PMID 30584557
- [Result] Tran KT, Nguyen PV, Dang TTU, Ton TNB. The Impacts of the High-Quality Workplace Relationships on Job Performance: A Perspective on Staff Nurses in Vietnam. Behav Sci (Basel). 2018 Nov 23;8(12):109. doi: 10.3390/bs8120109. PMID 30477199
- [Result] Wilson W, Raj JP, Narayan G, Ghiya M, Murty S, Joseph B. Quantifying Burnout among Emergency Medicine Professionals. J Emerg Trauma Shock. 2017 Oct-Dec;10(4):199-204. doi: 10.4103/JETS.JETS_36_17. PMID 29097859
- See also: An Analysis of Structure in Northern Cyprus Ministry of Health — http://www.tepav.org.tr/upload/files/1455007392-2.KKTC_Saglik_Bakanligi_Kurumsal_ve_Fonksiyonel_Analizi.pdf
- See also: Health Services Statistical Report in Northern Cyprus — http://saglik.gov.ct.tr/%C4%B0STAT%C4%B0ST%C4%B0K%C4%B0-B%C4%B0LG%C4%B0LER